CLINICAL TRIAL: NCT05994586
Title: The Effect of Mix AP029 on the Efficacy of Metformin Therapy and Its Side Effects in Patients With Type II Diabetes and on Mechanisms Related to Prediabetes in Patients With Impaired Carbohydrate-lipid Metabolism
Brief Title: The Efficacy of AP029 Mix in Patients With Impaired Carbohydrate Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AronPharma Sp. z o. o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 07-AP-MET
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Diabetes in Adolescence; PreDiabetes
Keywords: Type II diabetes; Prediabetes; Disorders of Carbohydrate Metabolism; Chokeberry; Elderberry
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AP029 mix - type II diabetes (Experimental): Patients with type II diabetes receiving metformin for up to 5 months
  Interventions: Dietary Supplement: AP029 mix
- AP029 mix - prediabetes (Experimental): Patients with pre-diabetic
  Interventions: Dietary Supplement: AP029 mix
- Placebo - type II diabetes (Placebo Comparator): Patients with type II diabetes receiving metformin for up to 5 months
  Interventions: Other: Placebo
- Placebo - prediabetes (Placebo Comparator): Patients with pre-diabetic
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: AP029 mix — Polyphenol-rich plant extracts Twice a day
  Arms: AP029 mix - prediabetes; AP029 mix - type II diabetes
Other: Placebo — Twice a day
  Arms: Placebo - prediabetes; Placebo - type II diabetes

SUMMARY:
The aim of the study is to demonstrate that a daily supplementation of AP029 Mix: I) has a positive effect on reducing side effects of metformin, while enhancing the therapeutic effect of metformin; II) normalizes prediabetes biomarkers in order to prevent further progression into diabetes.

DETAILED DESCRIPTION:
Randomized, double-blind, cross over study conducted under medical supervision on 1) group of 20 patients with type II diabetes and 2) group of 10 patients with prediabetes.

Study design: 2 months of AP029 supplementation, 1 month wash-out, 2 months of placebo intake. Patients will attend 4 visits. On each visit, the following parameters are analyzed: level of glucose, insulin, HbA1c, hsCRP lipid panel (total cholesterol (TC), triglycerides (TG), low density lipoprotein (LDL), HDL) and inflammatory and oxidative stress markers. In addition, a questionnaire of symptoms associated with metformin intake will be conducted

ELIGIBILITY:
Inclusion Criteria for type II diabetes:

* Women and men, 18-75 years old
* Patients diagnosed with type II diabetes mellitus
* Patients on metformin treatment up to 5 months
* BMI 20-35 kg/m2
* Signed informed consent

Inclusion Criteria for prediabetes:

* Women and men, 18-75 years old
* BMI 20-35 kg/m2
* Fasting blood glucose levels between 100 mg/dl and 125 mg/dl (5.6-6.9 mmol/l)
* Signed informed consent

Exclusion Criteria for type II diabetes:

* Patients diagnosed with type I diabetes
* Patients receiving insulin or other anti-diabetic medications
* Women who are pregnant, planning to become pregnant during the study, or breastfeeding
* Surgery within the last 6 months
* Intake of dietary supplements containing plant extracts rich in polyphenols and anthocyanins
* Intake of supplements containing: white mulberry, chromium, berberine
* Patients receiving glucocorticosteroids, immunosuppressants
* Oncological disease, autoimmune disease, severe liver dysfunction, tuberculosis, leukemia, multiple sclerosis, AIDS, rheumatoid arthritis, organ transplant
* Acute inflammation (C-reactive protein >20mg/dl)

Exclusion Criteria for prediabetes:

* Patients diagnosed with type I, II, LADA diabetes
* Patients receiving insulin or other anti-diabetic medications
* Women who are pregnant, planning to become pregnant during the study, or breastfeeding
* Surgery within the last 6 months
* Intake of dietary supplements containing plant extracts rich in polyphenols and anthocyanins
* Intake of supplements containing: white mulberry, chromium, berberine
* Patients receiving glucocorticosteroids, immunosuppressants
* Oncological disease, autoimmune disease, severe liver dysfunction, tuberculosis, leukemia, multiple sclerosis, AIDS, rheumatoid arthritis, organ transplant
* Acute inflammation (C-reactive protein >20mg/dl)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-11-26 (Estimated); Study Completion 2023-11-26 (Estimated)

PRIMARY OUTCOMES:
Glucose level | Baseline, 2 months, 3 months, 5 months
  Comparison of glucose level
Insulin level | Baseline, 2 months, 3 months, 5 months
  Comparison of insulin level
Discomfort related to metformin side effects | Baseline, 2 months, 3 months, 5 months
  Based on questionnaire

SECONDARY OUTCOMES:
Lipid panel (total cholesterol (TC), triglycerides (TG), low-density lipoprotein (LDL), HDL) | Baseline, 2 months, 3 months, 5 months
  Comparison of lipid panel markers
hsCRP level | Baseline, 2 months, 3 months, 5 months
  Comparison of hsCRP level
HbA1c level | Baseline, 2 months, 3 months, 5 months
  Comparison of hbA1c level

CONTACTS AND LOCATIONS:
Locations (1):
- Pomorskie Centrum Reumatologiczne im. dr Jadwigi Titz-Kosko, Sopot, Poland

IPD SHARING:
Plan to Share IPD: No